CLINICAL TRIAL: NCT04168840
Title: Ultrasound Parameters to Predict Difficult Airway
Status: Completed | Type: Observational
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Other Study IDs: UPDA
Record Dates: First submitted 2019-11-14; First posted 2019-11-19 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2020-01

CONDITIONS: Difficult Intubation
Keywords: ultrasound; difficult airway; difficult intubation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient undergoing general anesthesia with intubation: Patient undergoing general anesthesia with intubation We will explore clinical airway parameters and external ultrasound parameters of the airway
  Interventions: Diagnostic Test: Compare clinical test with ultrasound parameters

INTERVENTIONS:
Diagnostic Test: Compare clinical test with ultrasound parameters — Compare various clinical test with four ultrasound parameters to predict difficult intubation.

SUMMARY:
Ultrasound has become an essential tool for the daily work of any doctor, but in certain specialties such as Anaesthesiology, its use has greatly increased the safety offered to patients throughout the perioperative period, either to perform nerve blocks, for vascular access, intraoperative hemodynamic management or any other use that allows increasing quality of care.

The management of the upper airway and the diagnosis of pathological conditions are essential skills for any doctor especially for Anaesthesiologist, ER physician, or Intensive Care physician. Because an inadequate airway management continues to be an important contributor to patient mortality and morbidity, any tool that can improve it should be considered as an addition to conventional clinical evaluation.

Unfortunately, most of the clinical parameters that should allow us to assess a potential difficult airway, do not always lead us to an adequate prediction, that is why US(Ultrasound) is use as an emerging tool in many fields, is also gathering strength in this search for a definitive predictor parameter.

Ultrasound has many obvious advantages (safe,fast, repeatable, portable, widely available and gives dynamic images in real time).

Sonographic studies are operator-dependent and although the identification of basic structures could be acquired with only a few hours of training, but more complex studies require a learning curve of months or even years. The high frequency linear probe (5-14 MHz) is probably the most suitable for the airway because images are of superficial structures (within 0-5 cm below the skin surface).

The growing academic interest in the use of US to look for predictors of difficult airway is centred mainly on measurements at the level of pretracheal tissues.

But the greatest limitation of these studies is the disparity of the fat distribution that exists between different ethnic groups and and sexes, and the lack of standardization method in patient´s intubation conditions.

So, the investigator propose to assess different ultrasound windows at the level of pretracheal tissues such as independent predictors of Difficult Airway.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male or female) ASA I-III, aged between 18 and 90 years, undergoing scheduled surgery requiring orotracheal intubation. The signature of the informed consent is required authorizing its inclusion in the study.

Exclusion Criteria:

* Obesity class II defined as a BMI greater than 35.
* Pregnant.
* Cervical tumors, goiter or patients who have required radiotherapy at the cervical level
* Abnormalities that condition anatomy alterations such as facial / cervical fractures.
* Maxillofacial abnormalities
* People who cannot give their consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing scheduled surgery requiring orotracheal intubation.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
Anterior neck soft tissue thickness measured by ultrasound at hyoid bone | 5 minutes
  Distance from skin to the midline of hyoid bone measure with lineal ultrasound probe
Anterior neck soft tissue thickness measured by ultrasound at thyrohyoid membrane | 5 minutes
  Distance from skin to midline of epiglottis measure with lineal ultrasound probe
Anterior neck soft tissue thickness measured by ultrasound at anterior commissure of vocal cords | 5 minutes
  Distance from skin to anterior commisure of vocal cords measure with lineal ultrasound probe
Anterior neck soft tissue thickness measured by ultrasound at thyrohyoid membrane. Preepiglottic Area. | 5 minutes
  Calculated with distance from skin to midline of epiglottis and 1 centimeterto left and right side.

SECONDARY OUTCOMES:
Modified Mallampati Score | 1 minute
  Class I: Soft palate, uvula, fauces, pillars visible. Class II: Soft palate, major part of uvula, fauces visible. Class III: Soft palate, base of uvula visible. Class IV: Only hard palate visible. Class I is better than Class IV for not to be a difficult intubation.
Thyromental distance | 1 minute
  measured from the thyroid notch to the tip of the jaw with the head extended
Sternomental distance | 1 minute
  the distance from the suprasternal notch to the mentum and is measured with the head fully extended on the neck and the mouth closed
Interincisor distance | 1 minute
  DIstance in centimeters between fornt incisors
Upper Lip Bite Test | 1 minute
  upper lip bite criteria-class I = lower incisors can bite the upper lip above the vermilion line, class II = lower incisors can bite the upper lip below the vermilion line, and class III = lower incisors cannot bite the upper lip. Class I is the best for not to be a difficult intubation, class III means it´s posibble a difficult laryngoscopy.
neck circumference | 1 minute
  Using a flexible measuring tape in centimeters, neck circumference at the level of thethyroid cartilage will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Universidad de Navarra, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided